CLINICAL TRIAL: NCT00687778
Title: 11C-Acetate PET/CT Non-FDG-Avid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Einat Even-Sapir MD, PhD, Dept of Nuclear Medicine, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-EE-109-CTIL
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Soft Tissue Sarcomas; Thyroid Cancer; Lung Cancer; Indolent Lymphoma; Neuroendocrine Tumors; GIST; Uterine Malignancies; Carcinoma, Hepatocellular; Carcinoma, Lobular; Teratoma
Keywords: C11-Acetate; FDG; sarcoma; Measurement of C11-Acetate uptake in tumors which are often non-FDG avid.; Soft tissue sarcomas; well-differentiated thyroid cancer; well-differentiated and bronchoalveolar lung cancer; indolent lymphomas, neuroendocrine tumors; GIST; uterine malignancies; mucin-producing cancer; teratoma, hepatoma; HCC; lobular breast carcinoma
MeSH Terms: conditions — Sarcoma; Thyroid Neoplasms; Lung Neoplasms; Neuroendocrine Tumors; Carcinoma, Hepatocellular; Carcinoma, Lobular; Teratoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: 100 patients with newly diagnosed tumors, which are often non-FDG avid or show only low intensity uptake: Soft tissue sarcomas, well-differentiated thyroid cancer, well-differentiated and bronchoalveolar lung cancer, indolent lymphomas, neuroendocrine tumors, GIST, uterine malignancies, mucin-producing cancer, teratoma, hepatoma, HCC and lobular breast carcinoma.

SUMMARY:
F18-FDG is the widely used PET tracer in the routine practice of oncologic disease imaging using the technology of PET-CT. However, FDG-avidity is a characteristic of the individual tumor. There are various types of human malignancies, which are not taking FDG in access. In these cases FDG is not a sensitive tracer of imaging. In search for other tumor PET tracers, C11-Acetate has been shown recently in a few early studies to have a potential value in imaging of non-FDG-avid tumors.

The purpose of the current study is to assess the role of 11C-acetate PET in various tumors, which often are not detected by 18F-FDG and were not widely assessed until now.

DETAILED DESCRIPTION:
Recent publications have suggested the use of 11C-acetate as another PET tracer for tumor imaging. The accumulation of 11C-acetate in tumor cells is related to the highly active lipid metabolism in the cell membrane associated with tumor growth. 11C-acetate is channeled into the tricarboxylic acid cycle via acetyl coenzyme A and then incorporated via phosphatidylcholine into the cell membrane's phopholipids. Possible biochemical paths of acetate incorporation or accumulation include (a) entering the Krebs cycle from acetyl coenzyme A (acetyl CoA) or as an intermediate metabolite, (b) esterification to form acetyl CoA as a major precursor in ß-oxidation for fatty acid synthesis, (c) combining with glycine in heme synthesis, and (d) through citrate for cholesterol synthesis. Of all of these possible metabolic pathways, participation in free fatty acid (lipid) synthesis is believed to be the dominant method of incorporation in tumors.

The clinical data on the role of 11C-acetate PET in human tumors is being accumulated. Most clinical studies have investigated the role of 11C-acetate PET in detection of prostate cancer. 11C-acetate PET was found valuable in the detection of recurrent prostate cancer, both in the prostate bed, lymph nodes and distant metastases. The main advantage of 11C-acetate is that it does not show physiological accumulation in the urinary bladder as is the case with 18F -FDG and therefore may be appropriate for the detection of active pelvic disease.

Comparing the uptake of 18F-FDG and of 11C-acetate in patients with lung carcinoma, the latter was found superior in the identification of a bronchiolo-alveolar carcinoma which often show no intense FDG uptake.

In the case of hepatic masses, well-differentiated HCC tumors were detect by 11C-acetate while poorly differentiated types were detected by 18F-FDG.

These data suggest that 11C-acetate PET may be valuable in the detection of well-differentiation slow growing tumors and may have a complementary role to the routinely used 18F-FDG.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed tumors, which are often non-FDG avid or show only low intensity uptake:

  * Soft tissue sarcomas
  * well-differentiated thyroid cancer
  * well-differentiated and bronchoalveolar lung cancer
  * indolent lymphomas
  * neuroendocrine tumors
  * GIST
  * uterine malignancies
  * mucin-producing cancer
  * teratoma
  * hepatoma
  * HCC
  * lobular breast carcinoma
* Patients over the age of 18

Exclusion Criteria:

* patients under the age of 18 years
* pregnant and lactating women
* claustrophobic patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with newly diagnosed tumors, which are often non-FDG avid or show only low intensity uptake: Soft tissue sarcomas, well-differentiated thyroid cancer, well-differentiated and bronchoalveolar lung cancer, indolent lymphomas, neuroendocrine tumors, GIST, uterine malignancies, mucin-producing cancer, teratoma, hepatoma, HCC and lobular breast carcinoma.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Uptake of C11-Acetate and F18-FDG in tumor will be measured in SUV PET units | At completion of acuisition

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even-Sapir, MD, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Department of Nuclear Medicine, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel